CLINICAL TRIAL: NCT07232316
Title: Effect of Integrated Neuromuscular Inhibition Technique (INIT) Versus Conventional Exercise on Muscular Strength, Shoulder ROM and Scapular Deviation Among Young Adults With Scapular Dyskinesia II.
Brief Title: Effect of Integrated Neuromuscular Inhibition Technique on Scapular Dyskinesia Type 2
Acronym: INITonSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Syeda Sana Waheed, Principal Investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9050824SWPT; 9050824SWPT (Other: Ziauddin University)
Record Dates: First submitted 2025-09-23; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Scapular Dyskinesis
Keywords: scapular dyskinesis, shoulder rehabilitation, integrated neuromuscular inhibition technique

STUDY DESIGN:
Intervention Model Description: Group A: INIT group The practitioners first identified the latent trigger points to be treated within the using the palpation method and treated with ischemic pressure that the participant can tolerate. Pressure will be maintained at a participant-tolerated level, following standard ischemic compression procedures.. It will be continued until referred or local pain diminishes. This technique will be done for 90 secs and repeated 3 to 5 times After the ischemic compression therapist, the position of ease will be attained by maintaining the part of the desired muscle in the shortened position.
  MET is a soft tissue manipulation technique in which an individual actively performs muscle contraction in a controlled manner
  Group B receives conventional exercise that includes stretches and strengthening exercises of muscles involved in SD:
  For stretching: Should repeat 2-4 times increasing gradually with a 15-30 second hold.
  For strengthening: Active exercise for ten reps in 3 sets.
Who Masked: Participant
Masking Description: A simple random technique will be used with the envelope method for randomization.
  Two sets of envelopes entitled groups A and B will be presented to the participant before recruitment in the study so that 2 sets of envelopes are mutually exclusive and cannot be replaced in the set again.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A receives integrated neuromuscular inhibition technique. The total time commitment encompasses these assessment points spanning six weeks with each session lasting 45 minutes occurring three consecutive days a week.
  Interventions: Other: Intigrated Neuromuscular Inhibition Technique
- Group B (Experimental): Group B receives conventional exercise. The total time commitment encompasses these assessment points spanning six weeks with each session lasting 45 minutes occurring three consecutive days a week.
  Interventions: Other: Conventional Exercise

INTERVENTIONS:
Other: Intigrated Neuromuscular Inhibition Technique — The integrated Neuromuscular Inhibition Technique (INIT) combines ischemic compression, strain-counter strain, and muscle energy techniques.
  The practitioners first identified the latent trigger points to be treated using the palpation method and treated with ischemic pressure. This technique will be done for 90 seconds and repeated 3 to 5 times. After the ischemic compression therapist, the position of ease will be attained by maintaining the part of the desired muscle in the shortened position. It will be maintained for 20-30 sec. MET is a soft tissue manipulation technique in which an individual actively performs muscle contraction in a controlled manner. In this study, isometric contraction using post-isometric relaxation technique with stretching is used
  Arms: Group A
Other: Conventional Exercise — Group B receives conventional exercise that includes stretches and strengthening exercises of muscles involved in SD.
  For stretching: Should repeat 2-4 times increasing gradually with a 15-30 second hold.
  For strengthening: Active exercise for ten reps in 3 sets gradually increases for 15 reps in 3 stages. The intensity of exercise will be determined by the RM method using a yellow Thera band with an elastic range of 70%-80% that is i.50 kilograms per unit
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to learn whether the Integrated Neuromuscular Inhibition Technique (INIT) can influence shoulder motion, muscle strength, and scapular positioning in young adults with Scapular Dyskinesis Type II. This study will also compare INIT with a conventional exercise program.

The main questions the study aims to answer are:

* Does INIT affect shoulder range of motion compared with conventional exercise?
* Does INIT affect shoulder-girdle muscle strength?
* Does INIT influence scapular deviation as measured by a palpation meter? Participants will receive either INIT or conventional exercises three times per week for six weeks. Assessments will occur at baseline, week 4, and week 6 using a goniometer, dynamometer, and palpation meter. A physiotherapist that is the Principal Investigator and supervisor will monitor participants throughout the study.

DETAILED DESCRIPTION:
A total of 82 participants will be recruited using a multifaceted approach through pamphlets, emails, and WhatsApp groups. After enrollment, candidates will be screened by the principal investigator and re-evaluated by a clinical co-supervisor. Informed voluntary consent will be obtained before participation. Participants will be randomly allocated via the envelope method into:

* Treatment group: Integrated Neuromuscular Inhibition Technique (INIT)
* Control group: Conventional therapy Assessments will occur at baseline, week 4, and week 6 using a palpation meter (PALM), goniometer, and hand-held dynamometer. Each session will last 45 minutes and will be conducted three times per week for six weeks. The Scapular Assistance Test will be used initially to identify scapular dyskinesis, followed by PALM measurements-where positive values indicate upward and negative values indicate downward movement. The dynamometer will record peak force (Newtons) in a gravity-eliminated position. An orthopedic surgeon will monitor participant safety and manage any adverse events.

Integrated Neuromuscular Inhibition Technique (INIT):

INIT combines ischemic compression, strain-counter strain, and muscle energy technique (MET).

* Ischemic Compression: Latent trigger points in the upper trapezius, levator scapulae, rhomboids, and serratus anterior are palpated and compressed for 90 seconds, repeated 3-5 times based on participant tolerance.
* Strain-Counter Strain: The muscle is placed in a position of ease. For the upper trapezius and levator scapulae, the head is side-bent 10°-20° toward the affected side with the ipsilateral arm in abduction or flexion, held for 20-30 seconds.
* Muscle Energy Technique: Using post-isometric relaxation, participants perform gentle isometric contractions of the same muscles, followed by stretching.

Conventional Therapy (Control Group):

Participants perform stretching and strengthening for the same muscles.

* Stretching: Upper trapezius and levator scapulae-2-4 repetitions, holding 15-30 seconds each.
* Strengthening: Rhomboids and serratus anterior-10 repetitions × 3 sets, progressing to 15 repetitions × 3 sets using a yellow TheraBand (70-80% elasticity, approximately 1.5 kg/unit).

This six-week protocol will provide a standardized framework for comparing the two interventions using planned assessments

ELIGIBILITY:
Inclusion Criteria:

* ● Both male and female participants aged between 20-40 years will be diagnosed by an orthopedic consultant and screened by a physiotherapist through Scapular Assistant Test and a PALM meter.

  * Individuals presenting with scapular malposition and inferior medial border prominence, scapular dyskinesia type II with nonspecific symptoms.

Exclusion Criteria:

* Any diagnosed neurological deficit, i.e., hemiplegic limb, winged scapula due to lesions of the long thoracic or spinal accessory nerve.

  * Diagnosed Cervical related pathologies such as stenosis, myelopathy, and prolapsed intervertebral disk.
  * Diagnosed Shoulder-related pathology such as AC joint instability, rotator cuff pathology, history of shoulder surgery, and recent upper limb fracture.
  * Individual with neurovascular deficit and rib fracture.
  * Diagnosed chest deformity and scoliosis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Range of motion | Baseline
  The shoulder range of motion (flexion, abduction and external and internal rotation) will be using a goniometer with a reliability ICC=0.94.
Range of motion | 4 week
  The shoulder range of motion (flexion, abduction and external and internal rotation) will be using a goniometer with a reliability ICC=0.94.
Range of motion | 6 week
  Shoulder range of motion (flexion, abduction, and external and internal rotation) will be using a goniometer with a reliability ICC=0.94.
Muscular strength | Baseline
  The strength of spino scapular muscles will be measured by using hand-held dynamometer That measures peak isometric force generated by muscle groups with an inter-rater reliability ICC=0.98
Muscular strength | 4 week
  The strength of spino scapular muscles will be measured by using hand-held dynamometer That measures peak isometric force generated by muscle groups with an inter-rater reliability ICC=0.98
Muscular strength | 6 week
  The strength of spino scapular muscles will be measured by using hand-held dynamometer That measures peak isometric force generated by muscle groups with an inter-rater reliability ICC=0.98
Scapular deviation | Baseline
  PALM meter (performance Attainment Associate, St. Paul, MN, USA) will be used to measure Upward scapular deviation. It has calipers and an analogue inclinometer that can be used to calculate the horizontal distance between the scapula position and spine in scaption and coronal plane with an inter-rater reliability ICC=0.90-0.99
Scapular deviation | 4 week
  PALM meter (performance Attainment Associate, St. Paul, MN, USA) will be used to measure Upward scapular deviation. It has calipers and an analogue inclinometer that can be used to calculate the horizontal distance between the scapula position and spine in scaption and coronal plane with an inter-rater reliability ICC=0.90-0.99
Scapular deviation | 6 week
  PALM meter (performance Attainment Associate, St. Paul, MN, USA) will be used to measure Upward scapular deviation. It has calipers and an analogue inclinometer that can be used to calculate the horizontal distance between the scapula position and spine in scaption and coronal plane with an inter-rater reliability ICC=0.90-0.99

CONTACTS AND LOCATIONS:
Overall Officials: Amna Aamir Khan, PhD - PT, Study Director — Ziauddin University
Locations (1):
- Ziauddin University, College of Physical Therapy, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tang L, Chen K, Ma Y, Huang L, Liang J, Ma Y. Scapular stabilization exercise based on the type of scapular dyskinesis versus traditional rehabilitation training in the treatment of periarthritis of the shoulder: study protocol for a randomized controlled trial. Trials. 2021 Oct 18;22(1):713. doi: 10.1186/s13063-021-05654-2. PMID 34663424
- [Result] Roche SJ, Funk L, Sciascia A, Kibler WB. Scapular dyskinesis: the surgeon's perspective. Shoulder Elbow. 2015 Oct;7(4):289-97. doi: 10.1177/1758573215595949. Epub 2015 Jul 16. PMID 27582990
- [Result] Saadat Z, Hemmati L, Pirouzi S, Ataollahi M, Ali-Mohammadi F. Effects of Integrated Neuromuscular Inhibition Technique on pain threshold and pain intensity in patients with upper trapezius trigger points. J Bodyw Mov Ther. 2018 Oct;22(4):937-940. doi: 10.1016/j.jbmt.2018.01.002. Epub 2018 Jan 17. PMID 30368338
- [Result] Lytras D, Sykaras E, Christoulas K, Myrogiannis I, Kellis E. Effects of an integrated neuromuscular inhibition technique program on neck muscle strength and endurance in individuals with chronic mechanical neck pain. J Bodyw Mov Ther. 2019 Jul;23(3):643-651. doi: 10.1016/j.jbmt.2019.01.004. Epub 2019 Jan 28. PMID 31563383
- [Result] Saglam G, Telli H. The prevalence of scapular dyskinesia in patients with back, neck, and shoulder pain and the effect of this combination on pain and muscle shortness. Agri. 2022 Apr;34(2):100-108. doi: 10.14744/agri.2022.87059. PMID 35848815
- [Result] Kolber MJ, Hanney WJ. The reliability and concurrent validity of shoulder mobility measurements using a digital inclinometer and goniometer: a technical report. Int J Sports Phys Ther. 2012 Jun;7(3):306-13. PMID 22666645
- [Result] Kibler WB, Sciascia A. Evaluation and Management of Scapular Dyskinesis in Overhead Athletes. Curr Rev Musculoskelet Med. 2019 Dec;12(4):515-526. doi: 10.1007/s12178-019-09591-1. PMID 31760624
- [Result] Kheradmandi A, Kamali F, Ebrahimian M, Abbasi L. Comparison between dry needling plus manual therapy with manual therapy alone on pain and function in overhead athletes with scapular dyskinesia: A randomized clinical trial. J Bodyw Mov Ther. 2021 Apr;26:339-346. doi: 10.1016/j.jbmt.2020.11.017. Epub 2020 Nov 24. PMID 33992267
- [Result] Hickey D, Solvig V, Cavalheri V, Harrold M, Mckenna L. Scapular dyskinesis increases the risk of future shoulder pain by 43% in asymptomatic athletes: a systematic review and meta-analysis. Br J Sports Med. 2018 Jan;52(2):102-110. doi: 10.1136/bjsports-2017-097559. Epub 2017 Jul 22. PMID 28735288
- [Result] Gorji SM, Kazemi O, Shahrzad P, Marchetti PH. Efficacy of Six Weeks Stability Exercises on the Glenohumeral Joint of Female Tennis Players with Scapular Dyskinesia. Int J Exerc Sci. 2022 Jul 1;15(3):962-973. doi: 10.70252/RGVB2654. eCollection 2022. PMID 36158226
- [Result] Amorim CS, Gracitelli ME, Marques AP, Alves VL. Effectiveness of global postural reeducation compared to segmental exercises on function, pain, and quality of life of patients with scapular dyskinesis associated with neck pain: a preliminary clinical trial. J Manipulative Physiol Ther. 2014 Jul-Aug;37(6):441-7. doi: 10.1016/j.jmpt.2013.08.011. Epub 2014 Aug 3. PMID 25092553
- [Result] Chitale N Jr, Patil DS, Phansopkar P. Integrated Neuromuscular Inhibition Technique Versus Mulligan Mobilization on Functional Disability in Subjects With Nonspecific Low Back Pain: A Comparative Study. Cureus. 2022 Oct 13;14(10):e30253. doi: 10.7759/cureus.30253. eCollection 2022 Oct. PMID 36381847
- [Result] Okezue OC, Anamezie TH, Nene JJ, Okwudili JD. Work-Related Musculoskeletal Disorders among Office Workers in Higher Education Institutions: A Cross-Sectional Study. Ethiop J Health Sci. 2020 Sep;30(5):715-724. doi: 10.4314/ejhs.v30i5.10. PMID 33911832
- [Result] Baschung Pfister P, de Bruin ED, Sterkele I, Maurer B, de Bie RA, Knols RH. Manual muscle testing and hand-held dynamometry in people with inflammatory myopathy: An intra- and interrater reliability and validity study. PLoS One. 2018 Mar 29;13(3):e0194531. doi: 10.1371/journal.pone.0194531. eCollection 2018. PMID 29596450